CLINICAL TRIAL: NCT02034357
Title: Sleep Disordered Breathing and Its Impact on Neuro-cognitive Performance and Quality of Life in Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Parkinson Foundation (Other)
Responsible Party: Principal Investigator, Carlos Singer, Division Chief Parkinson Disease and Movement Disorders, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 20110265
Record Dates: First submitted 2013-12-15; First posted 2014-01-13 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Parkinson's Disease; Sleep Disordered Breathing; Sleep Obstructive Apnea
Keywords: Parkinson Disease; Sleep Disordered Breathing; Sleep Obstructive Apnea; Polysomnography; CPAP (continuous positive airway pressure) titration; CPAP (continuous positive airway pressure) treatment
MeSH Terms: conditions — Parkinson Disease; Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Microcephaly, Primary Autosomal Recessive, 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neurocognitive function (Other): Neurocognitive function assessment (verbal learning and memory) as measured by CVLT and sleep evaluations in Parkinson's disease patients at baseline, and after 4 months and 1 year of CPAP treatment
  Interventions: Other: Neurocognitive function; Other: Sleep evaluations

INTERVENTIONS:
Other: Neurocognitive function — Each eligible participant will complete a neuro-cognitive assessment as measured by CVLT at the beginning of the study. Neurocognitive evaluations will be repeated at 4-month and 1-year follow-up.
Other: Sleep evaluations — Each eligible participant will complete sleep questionnaires and undergo a baseline sleep study at the beginning of the study. The sleep questionnaires will be repeated at 4-month and 1-year follow-up.

SUMMARY:
The purpose of this study is to determine the impact of sleep and breathing problems during sleep on memory, attention, and general well being (quality of life) in people with Parkinson Disease.

DETAILED DESCRIPTION:
During the 2 year award period, we will prospectively enroll 200 patients with idiopathic Parkinson Disease (PD), who meet eligibility criteria below. All patients will undergo a baseline polysomnography (PSG) to diagnose Sleep Disordered Breathing (SDB) and will be asked to complete validated questionnaires to measure Sleep Quality, SDB risk, insomnia severity, daytime sleepiness, presence of restless leg syndrome (RLS), anxiety/depression, and quality of life. Medical records will be reviewed to determine co-morbidities and medication use. Each PD participant will undergo a full neurological examination, including the Unified Parkinson's Disease Rating Scale (UPDRS), the Hoehn & Yahr stage and a battery of neuro-cognitive measures at baseline. Patients with SDB will be offered PAP titration and treatment for 4 months. All patients (SDB [PAP compliant, non-compliant], and no SDB [controls]) will complete repeat neuro-cognitive evaluation, questionnaires, neurological evaluation and UPDRS assessment at 4 month and at 1 year follow-up. PD participants will be assessed in the "on" state in the morning. In the event that a participant goes "off" during testing, a break will be taken and participants will be given the option of taking their medication to return to the "on" state and resume testing or they can return later in the week to complete the evaluation. Although participants will understand the general purpose of the study, they will be blinded to the major study hypothesis. Neuropsychological examiners and the neurologist conducting the neurological exam will be blinded to the SDB status of the patient. Four month follow-up will be staggered according to enrolment date and will be completed by Year 2.

ELIGIBILITY:
Inclusion Criteria:

* Able to give consent.
* ≥18 years and have a Hoehn and Yahr stage at the time of enrollment of ≤3, clinical diagnosis of idiopathic Parkinson's Disease meeting the United Kingdom Parkinson's Disease Society Brain Bank criteria.
* Stable medical condition, including medications in the 1 month prior to enrollment.

Exclusion Criteria:

* Previous diagnosis of SDB with active use of Positive Airway Pressure (PAP), surgery for SDB or tracheostomy.
* Inability to read and comprehend English and/or Spanish at a grade 5 level.
* Prior history of neurosurgical procedures for PD or any other condition.
* Diagnosis of dementia as defined by Mini-mental state examination (MMSE) of < 26.
* History of major uncontrolled psychiatric illness.
* History of drug or alcohol abuse/dependence.
* History of major head injury or other neurological disease.
* Patients with observable craniofacial abnormalities that may be a relative contraindication to PAP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2011-06; Primary Completion 2013-08 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline Neurocognitive function in Parkinson's disease patients at 4 month and 1 year follow-up as measured by California Verbal Learning Test (CVLT) | Baseline, week 4, year 1
  Changes from Baseline Neurocognitive function (verbal learning and memory) in Parkinson's disease patients at 4 month and 1 year follow-up as measured by California Verbal Learning Test (CVLT).

SECONDARY OUTCOMES:
Prevalence of Sleep Disordered Breathing (SDB) in a diverse cohort of idiopathic PD patients. | Baseline
  Determine the Prevalence of Sleep Disordered Breathing (SDB) in a diverse cohort of idiopathic PD patients.
Prevalence of Insomnia in a diverse cohort of idiopathic PD patients. | Baseline
  Prevalence of Insomnia in a diverse cohort of idiopathic PD patients.
Prevalence of Poor Sleep Quality in a diverse cohort of idiopathic PD patients. | Baseline
  Prevalence of Poor Sleep Quality in a diverse cohort of idiopathic PD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Singer, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

REFERENCES:
- [Derived] Shafazand S, Wallace DM, Arheart KL, Vargas S, Luca CC, Moore H, Katzen H, Levin B, Singer C. Insomnia, Sleep Quality, and Quality of Life in Mild to Moderate Parkinson's Disease. Ann Am Thorac Soc. 2017 Mar;14(3):412-419. doi: 10.1513/AnnalsATS.201608-625OC. PMID 28231027